CLINICAL TRIAL: NCT06892405
Title: Using Ultrasound to Predict the Difficulty of Direct Laryngoscopy in Pediatrics.
Brief Title: Airway US in Predicting Difficult Pediatric Laryngoscopy
Acronym: AirwayUS
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Saad Abdel-Ghaffar, Professor of Anesthesia, intensive care and pain management, Assiut University
Other Study IDs: 04-2024-201007
Record Dates: First submitted 2025-03-21; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Airway Complication of Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: SonoSite™ S Series ultrasound — US measurements will be performed in the pre-operating room a
  , patients are placed in supine position with the head in a sniffing position on a surgical pillow and using the 15 MHz linear array transducer of the SonoSite™ S Series ultrasound in transverse position. A scan is made from the skin surface of the floor of the mouth to the trachea exerting the minimum possible pressure to identify the structures correctly.
  Other Names: US

SUMMARY:
The hypothesis of this study is that ultrasound measurements may improve the preoperative detection of difficult laryngoscopy (DL) in pediatrics. The primary objective of this study will be to evaluate the usefulness for the prediction of a DL of five ultrasound measurements obtained from the neck skin to three structures of the upper airway (hyoid, epiglottis and anterior commissure of the vocal cords). Secondary objectives will include establishing, if possible, a cut-off point in these measurements; to compare these measures against the classic pre-intubation clinical screening tests.

DETAILED DESCRIPTION:
Current advances in airway management training have reduced the risk associated with an unanticipated DL but have not been able to reduce its incidence in clinical practice. The addition of new video laryngoscopes in our clinical practice seems to offer a paradigm shift to face a DL with promising results. However, theses authors also indicated that expertise in video laryngoscopy requires prolonged training and practice. Otherwise, a growing number of publications have showed that some ultrasound measurements may improve our anticipation of a DL because of its high accuracy to offer detailed anatomical images of the airway, absence of ionizing radiations, accessibility and reproducibility. Among all the ultrasound parameters studied, distance from skin to epiglottis with a cut-off point of 2.10 cm, showed the best predictive ability with a sensitivity of 83.33%3 and a specificity of 73.33%, for predicting difficulty in airway management in routine clinical practice. The aim of this study is to investigate the efficacy of US-measured airway structures in predicting difficult laryngoscopy (defined as CL grade III and IV).

ELIGIBILITY:
Inclusion Criteria:

* Gender both males and females
* ASA Class I and II
* Age 2 years to 6
* Children scheduled for elective surgery under general anesthesia requiring orotracheal intubation after classical laryngoscopy.

Exclusion Criteria:

* Congenital upper airway malformation,
* Head and neck swellings,
* Scars,
* Radiation to the neck,
* Tracheotomy,

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 2-6 years, ASA I, II who will be scheduled for elective surgery under general anesthesia requiring orotracheal intubation after classical laryngoscopy.
Sampling Method: Probability Sample
Enrollment: 49 (Estimated)
Dates: Start 2025-04-20 (Estimated); Primary Completion 2027-04-20 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
prediction of a Difficult laryngoscopy of five ultrasound measurements obtained from the neck skin to three structures of the upper airway (hyoid, epiglottis and anterior commissure of the vocal cords). | Preoperative
  To evaluate the accuracy of five ultrasound measurements obtained from the neck skin to three structures of the upper airway (hyoid, epiglottis and anterior commissure of the vocal cords). Namely the DSH, DSE, DSG, DSH+DSE, and DSH-DSE in prediction of difficult laryngoscopy.

SECONDARY OUTCOMES:
The Modified Mallampati Score (MMS). | At Intubation
  The Modified Mallampati Score (MMS):
  * Class I: Soft palate, uvula, fauces, pillars visible.
  * Class II: Soft palate, major part of uvula, fauces visible.
  * Class III: Soft palate, base of uvula visible.
  * Class IV: Only hard palate visible.
The thyromental distance (TMD) | preoperative
  The thyromental distance (TMD) is the distance from the chin (mentum) to the top of the notch of the thyroid cartilage with the head fully extended measured by a ruler.
The upper lip bite test (ULBT) | Preoperative
  The upper lip bite test (ULBT) performed by an anesthesiologist associated with this research and a specialist with more than 10 years of experience and in charge of the operating room.

CONTACTS AND LOCATIONS:
Overall Officials: Hala S Abdel-Ghaffar, MD, Principal Investigator — Assiut University
Locations (1):
- Assiut university Pediatric hospital, Asyut, Assiut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No